CLINICAL TRIAL: NCT03316690
Title: The Interaction Between Metformin and Physical Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristian Karstoft (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Kristian Karstoft, Principal Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-17012307
Record Dates: First submitted 2017-10-03; First posted 2017-10-20 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Impaired Glucose Tolerance; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin treatment (Experimental)
  Interventions: Drug: Metformin treatment; Behavioral: Physical training
- Placebo treatment (Placebo Comparator)
  Interventions: Drug: Placebo treatment; Behavioral: Physical training

INTERVENTIONS:
Drug: Metformin treatment — Daily treatment with metformin tablets for 101 days according to the following scheme:
  Day 1-4: Metformin tablet 500 mg x 2 Day 5-8: Metformin tablet 1000 + 500 mg Day 9-101: Metformin tablet 1000 mg x 2
  Arms: Metformin treatment
Drug: Placebo treatment — Daily treatment with placebo tablets for 101 days according to the following scheme:
  Day 1-4: Placebo tablet 500 mg x 2 Day 5-8: Placebo tablet 1000 + 500 mg Day 9-101: Placebo tablet 1000 mg x 2
  Arms: Placebo treatment
Behavioral: Physical training — Twelve weeks of supervised physical training (4 times per week, 45 min per session, mean intensity at 70% of maximal oxygen consumption rate)

SUMMARY:
Physical activity is a first line treatment for patients with type 2 diabetes (T2D), however, the vast majority of patients with T2D do not achieve satisfying glycemic control with physical activity alone, which is why pharmacological treatment with metformin is most often initiated.

It is known that metformin and exercise both activates 5' adenosine monophosphate-activated protein kinase (AMPK) in skeletal muscle and liver, and the activation of AMPK results in many different metabolic effects, including improvements in glycemic control. Because of this similarity in mechanism of action, an interaction between metformin and exercise is plausible, but knowledge in the area is sparse. Thus, the aim of this study is to assess the effects of training with and without concomitant metformin treatment, in order to investigate whether an interaction between the two occur.

Subjects with impaired glucose tolerance will all undergo 12 weeks of training but will be randomized (1:1) to concomitant metformin/placebo treatment in a double-blinded way. Experimental days will be performed before randomisation (before initiation of metformin/placebo treatment), before initiation of the training period and after the training period.

ELIGIBILITY:
Inclusion Criteria:

* Glucose-lowering-medication naïve T2D and/or subjects with impaired glucose tolerance defined as: 2-h plasma glucose (PG) in the 75-g OGTT (7.8-11.0 mmol/L) and/or HbA1c (39-47 mmol/mol)
* Caucasian
* BMI > 25 but < 40 kg/m2
* Low to moderate physically active (≤90 min of structured physical activity/week)

Exclusion Criteria:

* Pregnancy
* Smoking
* Glucose-lowering treatment
* Treatment with steroids and other immunomodulating drugs
* Contraindication to increased levels of physical activity
* Liver disease (ALAT elevated more than 3 times above upper normal limit, or reduce levels of the liver function markers albumin and KF II+VII+X)
* Renal insufficiency (eGFR<60 ml/min)
* Prior history of lactic acidosis
* HbA1c >55 mmol/mol and/or 2-hPG in the 75-g OGTT > 15 mmol/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change in postprandial glycemic control as assessed by mean blood glucose concentration during a 4 hour mixed-meal tolerance test | Day 0 (before randomisation), 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)

SECONDARY OUTCOMES:
Change in free-living glycemic control | Day 0 (before randomisation), 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
  Blood HbA1c levels
Change in endogenous glucose production as assessed by rate of infused glucose tracer appearance in blood | Day 0 (before randomisation), 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
Change in exogenous glucose uptake as assessed by rate of ingested glucose tracer appearance in blood | Day 0 (before randomisation), 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
Change in peripheral glucose uptake as assessed by rate of glucose disappearance from blood | Day 0 (before randomisation), 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
Change in maximal oxygen consumption | Day 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
  Maximal oxygen uptake during an incremental bicycle test
Change in body weight | Day 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
  Body weight measured by standard procedures
Change in lean body mass | Day 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
  Lean body mass evaluated via Dual energy x-ray absorptiometry (Dxa)
Change in total fat mass | Day 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
  Total body fat mass evaluated via Dual energy x-ray absorptiometry (Dxa)
Change in visceral fat mass | Day 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
  Visceral fat mass evaluated via magnetic resonance imaging (MRI) scans
Change in AMPK activity in skeletal muscle | Day 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
  AMPK activity measured via western blotting and activity assays
Change in skeletal muscle oxidative stress | Day 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
  Muscle mitochondrial oxidative stress measured via respirometry in muscle biopsies
Change in systemic oxidative stress | Day 0 (before randomisation), 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
  Systemic oxidative stress measured via RNA/DNA oxidation products in urine
Maximal mitochondrial respiration | Day 17 (after initiation of metformin/placebo treatment), 101 (after 12 weeks of training)
  Maximal mitochondrial respiration measured via respirometry in muscle biopsies
Training heart rate | Average heart rate during all training sessions (through study completion, [Day 101])
  Heart rate will be measured continuously during all training sessions
Training rate of perceived exertion | Average rate of perceived exertion of all training sessions (through study completion, [Day 101])
  Rate of perceived exertion measured via a Borg scale (range 6-20 where higher values indicate higher rate of perceived exertion) will be assessed for each training session

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Karstoft, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Center for aktiv sundhed, Copenhagen, Copenhagen N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pilmark NS, Oberholzer L, Halling JF, Kristensen JM, Bonding CP, Elkjaer I, Lyngbaek M, Elster G, Siebenmann C, Holm NFR, Birk JB, Larsen EL, Lundby AM, Wojtaszewski J, Pilegaard H, Poulsen HE, Pedersen BK, Hansen KB, Karstoft K. Skeletal muscle adaptations to exercise are not influenced by metformin treatment in humans: secondary analyses of 2 randomized, clinical trials. Appl Physiol Nutr Metab. 2022 Mar;47(3):309-320. doi: 10.1139/apnm-2021-0194. Epub 2021 Nov 16. PMID 34784247
- [Derived] Pilmark NS, Lyngbaek M, Oberholzer L, Elkjaer I, Petersen-Bonding C, Kofoed K, Siebenmann C, Kellenberger K, van Hall G, Abildgaard J, Ellingsgaard H, Lauridsen C, Ried-Larsen M, Pedersen BK, Hansen KB, Karstoft K. The interaction between metformin and physical activity on postprandial glucose and glucose kinetics: a randomised, clinical trial. Diabetologia. 2021 Feb;64(2):397-409. doi: 10.1007/s00125-020-05282-6. Epub 2020 Sep 26. PMID 32979074